CLINICAL TRIAL: NCT01381159
Title: Motivational Intervention for Asthma Control Trial
Brief Title: Motivational Intervention for Asthma
Acronym: MI-ACT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal (Other)
Collaborators: Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Simon Bacon, Researcher, Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MBMC002; MOP 111123 (Other Grant/Funding Number: Canadian Institutes of Health Research)
Record Dates: First submitted 2011-06-21; First posted 2011-06-27 (Estimated); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Asthma
Keywords: Adherence; Asthma Control; Asthma Quality Of Life; Motivational Communication; Motivational Interviewing
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Motivational Communication (Experimental): Up to 3 x 30 minute brief MC sessions within 4-6 week period
  Interventions: Behavioral: Motivational Communication
- Control (Placebo Comparator): Usual care
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Motivational Communication — Brief MC sessions focused on medication adherence within 4-6 week period
  Arms: Motivational Communication
Behavioral: Control — Standard medical care
  Arms: Control

SUMMARY:
The high burden of asthma appears to be related to poor asthma control, which is associated with more frequent asthma symptoms, greater bronchodilator use and functional impairment, and worse pulmonary function. Despite the availability of effective treatments, more than 58% of asthmatics are poorly controlled. Daily adherence to inhaled corticosteroid (ICS) regimens is considered by experts to be one of the most important behavioural factors linked to achieving optimal asthma control. However, there is a paucity of research on interventions specifically designed to improve ICS adherence among adult asthmatics. The vast majority of intervention studies to date used atheoretical interventions to target behaviour change, relying mainly upon educational approaches which have been criticised for "failing to translate knowledge into action." This may be due to the fact that most education-based approaches do not specifically address or help patients overcome ambivalence about behaviour change, which is necessary for ensuring daily adherence. Motivational communication (MC) is a client-centred intervention that focuses on enhancing intrinsic motivation to change a particular behaviour, and exploring and resolving ambivalence about behaviour change. Brief MC sessions (e.g., 1-5 x 15-30 minute sessions) have been shown to improve a variety of health behaviours (e.g., reduce alcohol consumption, improve dietary habits, increase exercise behaviour, and improve medication adherence) and health outcomes (reduce blood pressure, body mass index, and cholesterol levels). However, no studies to date have assessed the efficacy of using MC to improve ICS adherence in asthmatics. This study aims to assess the efficacy of using MC to improve daily medication (ICS) adherence in a sample of poorly controlled, non-adherent asthmatics. It is hypothesized that patients randomized to the MC condition will exhibit significantly improved ICS adherence at 6 and 12-months post-intervention, independent of baseline levels and covariates, relative to patients randomized to the usual care control condition.

DETAILED DESCRIPTION:
Background: The high burden of asthma, which affects 300 million people worldwide, appears to be related to poor asthma control, which is associated with more frequent asthma symptoms, greater bronchodilator use and functional impairment, and worse pulmonary function. The availability of effective treatments suggests that asthma can be well controlled in most patients. However, Canadian statistics reveal that over 58% of asthmatics are poorly controlled. Achieving optimal asthma control relies upon several behavioral factors, including minimizing exposure to known triggers (e.g., pets, dust, pollen) and improving health behaviors (e.g,. quitting smoking and adhering to medication). Of these, daily adherence to inhaled corticosteroid (ICS) regimens is considered by experts to be one of the most important behavioral factors linked to achieving optimal asthma control. This is because taking ICS medications as prescribed (i.e., good adherence) has been shown to be effective for achieving good asthma control even in patients who fail to adequately manage/minimize exposure to known triggers (e.g., indoor allergens, exercise). Despite the efficacy of ICS's, recent trends in adherence behaviour suggest that asthmatics are not adherent to these medications, with rates being as low as 32%, even in patients with severe asthma. Explanations range from simply forgetting to having distorted/ erroneous illness and medication beliefs. Currently, there is a paucity of research on interventions specifically designed to improve ICS adherence among adult asthmatics. Most previous work has been conducted in pediatric samples which have yielded inconsistent results that are difficult to generalize to adult samples. Of the studies conducted among adults, most suffer from important methodological limitations (e.g., small sample sizes, no intent to treat analyses, failure to control for contact time, no objective measure of adherence) that make it difficult to either generalize findings or interpret them with confidence. Most importantly, the vast majority of intervention studies to date used atheoretical interventions to target behaviour change, relying mainly upon educational approaches which have been criticised for "failing to translate knowledge into action." This may be due to the fact that most education-based approaches do not specifically address or help patients overcome ambivalence about behaviour change, which is necessary for ensuring daily adherence. Motivational communication (MC) is a client-centred intervention that focuses on enhancing intrinsic motivation to change a particular behaviour (i.e., take medication as prescribed), and exploring and resolving ambivalence about behaviour change. Brief MC sessions (e.g., 1-5 x 15-30 minute sessions) have been shown to improve a variety of health behaviours (e.g., reduce alcohol consumption, improve dietary habits, increase exercise behaviour, and improve medication adherence) and health outcomes (reduce blood pressure, body mass index, and cholesterol levels). No studies to date have assessed the efficacy of using MC to improve ICS adherence in asthmatics. Objective: The purpose of this study is to conduct a single site RCT to assess the efficacy of using MC to improve daily medication (ICS) adherence in a sample of poorly controlled, non-adherent asthmatics. A brief (3-5 x 15-30 minute sessions), manualized MC intervention was developed by our laboratory using pilot funding. This intervention is empirically-driven and uses established behavioural and motivational strategies to encourage change. Methods: 182 poorly controlled, non-adherent adult asthmatics will be recruited from the outpatient asthma clinic of Hôpital du Sacré-Coeur de Montreal (HSCM). Patients will be screened on the day of their asthma clinic visit to verify eligibility. Eligible patients consenting to have their medical and pharmacy records verified by the research team and who are identified as both having poorly controlled asthma (Asthma Control Questionnaire score ≥1.25) and being non-adherent to ICS medication (filled < 50% of their ICS medication in the last year) will be invited to participate in the study. Patients will undergo baseline assessments (pulmonary function, asthma control, self-efficacy, and quality of life) and will then be randomly assigned to a usual care + MC or usual care comparison group. This trial has been designed to conform to the CONSORT guidelines. The primary outcome measure will be ICS adherence at 12 months post-intervention, with preliminary analyses conducted at 6-months post-intervention. Adherence will be measured according to the following validated equation: # of treatment days (based on the # of canisters filled at the pharmacy x the duration of each prescription) divided by the # of prescription days (# of days the patient is expected to be taking his/her medication). Data will be obtained by accessing the patient's pharmacy records and drug insurance databases (i.e., RAMQ, reMed). Secondary outcomes include self-reported medication adherence, adherence motivation, stage of change, pulmonary function, asthma control, self-efficacy, and quality of life scores 6 & 12 months post-intervention. Impact: This will be the first appropriately designed RCT to test the impact of a brief, manualized MC intervention on asthma medication (ICS) adherence that may be easily incorporated into existing education programs and/or clinical practice and may significantly improve asthma outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years and older
* Primary diagnosis of moderate-severe persistent asthma (as per GINA)
* Prescribed inhaled corticosteroid medication (min dose of 250 µg fluticasone equivalent per day) for at least 12 consecutive months
* Uncontrolled asthma (≥ 1.25 on the Asthma Control Questionnaire)
* Covered by a drug insurance plan (e.g., RAMQ)
* Non-adherent to ICS medication (based on having filled less than 50% of their prescriptions over the last year)
* Able to speak English or French.

Exclusion Criteria:

* Any other medical condition that confers greater illness morbidity than asthma (e.g., active cancer)
* Severe psychopathology (e.g., schizophrenia)
* Apparent cognitive or language deficit
* Are or plan to become pregnant or move outside of Quebec over the course of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2019-08 (Actual); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Inhaled corticosteroid adherence | 12 months post-intervention
  Inhaled corticosteroid adherence measured according to the following validated equation: # of treatment days (based on the # of canisters filled at the pharmacy x the duration of each prescription) divided by the # of prescription days (# of days the patient is expected to be taking his/her medication)

SECONDARY OUTCOMES:
Inhaled corticosteroid adherence | 6 months post-intervention
  Inhaled corticosteroid adherence measured according to the following validated equation: # of treatment days (based on the # of canisters filled at the pharmacy x the duration of each prescription) divided by the # of prescription days (# of days the patient is expected to be taking his/her medication)
Asthma Control Questionnaire (Juniper) | 12 months post-intervention
  Self report measure of asthma symptoms
Asthma Control Test | 12 months post-intervention
  Self report measures of asthma symptoms
Asthma Self-Efficacy Scale (Tobin) | 12 months post-intervention
  Self report measure of asthma self-efficacy, i.e., perceived ability to deal with asthma
Mini Asthma Quality of Life Questionnaire (Juniper) | 12 months post-intervention
  Self report measure of how asthma influences quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Kim L Lavoie, PhD, Principal Investigator — Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal; Simon L Bacon, PhD, Study Chair — Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal
Locations (1):
- Hopital du Sacre-Coeur de Montreal, Montreal, Quebec, Canada

REFERENCES:
- See also: Website of the research lab — http://mbmc-cmcm.ca